CLINICAL TRIAL: NCT01126528
Title: The Effect of Antenatal Vitamin D Supplementation on Maternal-fetal Vitamin D Status and Neonatal Immune Function: a Randomized Controlled Trial in Bangladesh
Brief Title: Antenatal Vitamin D3 Supplementation in Bangladesh: Randomized Controlled Trial
Acronym: AViDD-2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Responsible Party: Principal Investigator, Abdullah Baqui, Professor, Johns Hopkins Bloomberg School of Public Health
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: JHU-IRB2481; 02829-5 (Other Grant/Funding Number: Thrasher Research Fund)
Record Dates: First submitted 2010-05-18; First posted 2010-05-19 (Estimated); Last update posted 2012-08-17 (Estimated); Status verified 2012-08

CONDITIONS: Pregnancy
Keywords: Vitamin D; cholecalciferol; Micronutrients; Developing countries; Bangladesh; Infant, Newborn; Reproductive Health; Infant, Newborn, Diseases; Perinatology; Immunology; cathelicidin; Maternal Nutrition Physiology
MeSH Terms: conditions — Infant, Newborn, Diseases | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vitamin D3 (Experimental): Vitamin D3 (cholecalciferol)
  Interventions: Dietary Supplement: Vitamin D3
- Control (Placebo Comparator): Placebo control group
  Interventions: Dietary Supplement: Placebo control

INTERVENTIONS:
Dietary Supplement: Vitamin D3 — 35,000 IU per week, started at 26-29 weeks gestation, until delivery.
  Other Names: Cholecalciferol; Vigantol Oil
  Arms: Vitamin D3
Dietary Supplement: Placebo control — Miglyol 812, administered weekly from 26-29 weeks gestation until delivery.
  Arms: Control

SUMMARY:
This study is a randomized placebo-controlled trial of oral weekly vitamin D3 (cholecalciferol) supplementation during the third trimester of pregnancy among women in Dhaka, Bangladesh. The overall goal of the study is to establish whether there is evidence that improving vitamin D status among pregnant women in Bangladesh will enhance the resistance of the infant offspring to infection.

The aims of the study are to assess the effect of supplementation on 1) maternal and infant vitamin D status (based on blood concentrations of a vitamin D metabolite) and, 2) markers of neonatal immune function.

DETAILED DESCRIPTION:
The primary aims of this study are:

AIM #1 - To assess the effect of weekly antenatal administration of oral vitamin D3 (875 mcg/week = 35,000 IU week ≈ 5,000 IU per day) started in the third trimester (26-29 weeks gestation) on maternal vitamin D status and fetal-neonatal vitamin D status (cord blood), in comparison to a placebo control supplement.

AIM #2 - To demonstrate the maternal and fetal safety of weekly maternal antenatal (second and third-trimester) vitamin D supplementation at a dose of 875 mcg/week by monitoring maternal serum calcium, urinary calcium excretion, cord blood calcium concentration, and newborn clinical parameters.

AIM #3 - To measure the effect of antenatal vitamin D supplementation on selected biomarkers of fetal-neonatal immune function in cord blood: in vitro stimulated cord blood mononuclear cell (CBMC) LL-37 expression, gene expression related to inflammatory and immunoregulatory pathways, Th1/Th2 cytokine secretion, and bactericidal properties.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 to <35 years.
* Current residence in Dhaka at a fixed address
* Plans to have the delivery performed at the Shimantik maternity center, and to stay in Dhaka throughout the pregnancy and for at least one month past the date of delivery.
* Gestational age of 26th to 29th (inclusive), estimated based on the first day of the last menstrual period (LMP).

Exclusion Criteria:

* Use of any dietary supplement containing more than 400 IU/day (10 mcg/day) of vitamin D within the month prior to enrolment, or refusal to stop taking supplemental vitamin D at any dose after enrollment.
* Current use of anti-convulsant or anti-mycobacterial (tuberculosis) medications.
* Severe anemia (hemoglobin concentration < 70 g/L).
* Complicated medical or obstetric history that may increase the risk of preterm birth or labor/delivery complications, based on self-report or clinical assessment by physician (e.g., cardiovascular disease, uterine hemorrhage, placenta previa, threatened abortion, hypertension, preeclampsia, preterm labor, or multiple gestation).
* Prior history of delivery of an infant with a major congenital anomaly, birth asphyxia, or perinatal death (stillbirth or death within first week of life).

Ages: 18 Years to 34 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 160 (Actual)
Dates: Start 2010-08; Primary Completion 2011-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Serum 25-hydroxyvitamin D concentration | Maternal: during 3rd trimester; Neonatal (cord blood)
  Biomarker of vitamin D status.

SECONDARY OUTCOMES:
Serum calcium concentration | Maternal:3rd trimester; Cord blood.
Urine Ca:Cr ration | Maternal- 3rd trimester
Neonatal immune function | Cord blood
  Selected markers of innate and adaptive immunity.
Infant growth | Postnatal observational follow-up phase
  Infant growth parameters during postnatal follow-up, up to 12 months of age
Infant and maternal postnatal vitamin D status | Postnatal observational follow-up phase
Neonatal serum calcium | 1st week postnatal
  Infant serum calcium during the first week postnatal.

CONTACTS AND LOCATIONS:
Overall Officials: Abdullah Baqui, MBBS, Principal Investigator — JHSPH; ICDDR,B; Daniel Roth, MD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health; Rubhana Raqib, PhD, Principal Investigator — International Centre for Diarrhoeal Disease Research, Bangladesh
Locations (1):
- International Centre for Diarrheal Disease Research, Bangladesh (ICDDR,B), Dhaka, Dhaka Division, Bangladesh

REFERENCES:
- [Derived] Palacios C, Kostiuk LL, Cuthbert A, Weeks J. Vitamin D supplementation for women during pregnancy. Cochrane Database Syst Rev. 2024 Jul 30;7(7):CD008873. doi: 10.1002/14651858.CD008873.pub5. PMID 39077939
- [Derived] Akhtar E, Mily A, Haq A, Al-Mahmud A, El-Arifeen S, Hel Baqui A, Roth DE, Raqib R. Prenatal high-dose vitamin D3 supplementation has balanced effects on cord blood Th1 and Th2 responses. Nutr J. 2016 Aug 9;15(1):75. doi: 10.1186/s12937-016-0194-5. PMID 27506771
- [Derived] Harrington J, Perumal N, Al Mahmud A, Baqui A, Roth DE. Vitamin D and fetal-neonatal calcium homeostasis: findings from a randomized controlled trial of high-dose antenatal vitamin D supplementation. Pediatr Res. 2014 Sep;76(3):302-9. doi: 10.1038/pr.2014.83. Epub 2014 Jun 17. PMID 24937546
- [Derived] Roth DE, Perumal N, Al Mahmud A, Baqui AH. Maternal vitamin D3 supplementation during the third trimester of pregnancy: effects on infant growth in a longitudinal follow-up study in Bangladesh. J Pediatr. 2013 Dec;163(6):1605-1611.e3. doi: 10.1016/j.jpeds.2013.07.030. Epub 2013 Aug 30. PMID 23998516
- [Derived] Roth DE, Al Mahmud A, Raqib R, Akhtar E, Perumal N, Pezzack B, Baqui AH. Randomized placebo-controlled trial of high-dose prenatal third-trimester vitamin D3 supplementation in Bangladesh: the AViDD trial. Nutr J. 2013 Apr 12;12:47. doi: 10.1186/1475-2891-12-47. PMID 23587190